CLINICAL TRIAL: NCT06442124
Title: The Effect of BMI on Gluteus Maximum Activity in Adulthood With Sacroiliac Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy, Ahram Canadian University
Other Study IDs: P.T-REC-012/005149
Record Dates: First submitted 2024-05-13; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sacroiliac Joint Dysfunction; Obesity; EMG
MeSH Terms: conditions — Obesity | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (A):: o Group (A): will includes subjects with sacroiliac dysfunction and their body mass index < 25
  Interventions: Diagnostic Test: Electromyography (EMG)
- Group (B):: o Group (B): will includes subjects with sacroiliac dysfunction and their body mass index > 25.
  Interventions: Diagnostic Test: Electromyography (EMG)

INTERVENTIONS:
Diagnostic Test: Electromyography (EMG) — The present study will be conducted to add a new information to the body of knowledge of physical therapy profession as it will investigate the effect of BMI on gluteus maximum activity recorded by EMG in adulthood with sacroiliac dysfunction

SUMMARY:
PURPOSE:

This study will be conducted to investigate the effect of BMI on gluteus maximum activity in adulthood with sacroiliac dysfunction BACKGROUND: Sacroiliac joint (SIJ) pain is pain arising from SIJ structures and SIJ dysfunction (SIJD) generally refers to aberrant position or movement of SIJ structures . An estimated 15-30% of all low back pain cases are due to SIJ pain The present study will be conducted to add a new information to the body of knowledge of physical therapy profession as it will investigate the effect of BMI on gluteus maximum activity in adulthood with sacroiliac dysfunction

HYPOTHESES:

. •There will be no effect of BMI on gluteus maximum activity in adulthood with sacroiliac dysfunction

RESEARCH QUESTION:

* Do BMI has an effect on gluteus maximum activity in adulthood with sacroiliac dysfunction?

ELIGIBILITY:
Inclusion Criteria:

- adulthood with sacroiliac dysfunction

* Their ages will range from 20-40 years old.
* Their BMI will be less than 20- 30kg/m2.
* All of them suffer from mild to moderate degree of sacroiliac pain.
* The subjects complain from sacroiliac pain for 1 month ago

Exclusion Criteria:

* Exclusion criteria were a history of any of the following condition:

  * inflammatory diseases or any rheumatic disorders,
  * a history of vertebral fractures
  * surgical spinal fixation.
  * •any neurological disorders like MS

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects:
  A total of 60 male & female subjects, diagnosed with sacroiliac dysfunction participated in this study. Their BMI will from 20- 30kg/m2.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
gluteus maximum muscle activity measured by Electromyography (EMG) | up to 8 weeks
weight and height will be combined to report BMI in kg/m^2) | up to 8 weeks
visual analogue scale for pain | up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Canadian university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No